CLINICAL TRIAL: NCT03981952
Title: Phase 1 Randomized, Placebo-Controlled, Dose-Escalation Study of the Safety, Reactogenicity, and Immunogenicity of Trivalent (S. Enteritidis/S. Typhimurium/S. Typhi Vi) Conjugate Vaccine Against Invasive Salmonella Disease Administered Parenterally to Healthy U.S. Adults
Brief Title: Salmonella Conjugates CVD 1000: Study of Responses to Vaccination With Trivalent Invasive Salmonella Disease Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Wilbur Chen, MD, MS, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00084998
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Step 1) (Experimental): Individuals receive one dose of either 6.25 µg of the trivalent vaccine or placebo. Subsequent blood samples are taken for immunological testing.
  Interventions: Biological: Trivalent Invasive Salmonella Disease Vaccine (6.25 µg); Other: Placebo
- Cohort B (Step 2) (Experimental): Individuals receive one dose of either 12.5 µg of the trivalent vaccine or placebo. Subsequent blood samples are taken for immunological testing.
  Interventions: Biological: Trivalent Invasive Salmonella Disease Vaccine (12 µg); Other: Placebo
- Cohort C (Step 3) (Experimental): Individuals receive one dose of either 25 µg of the trivalent vaccine or placebo. Subsequent blood samples are taken for immunological testing.
  Interventions: Biological: Trivalent Invasive Salmonella Disease Vaccine (25 µg); Other: Placebo
- Cohort D (Experimental): Individuals receive one or two doses of the highest, well-tolerate dose among Cohorts A-C of the trivalent vaccine or placebo. Subsequent blood samples are taken for immunological testing.
  Interventions: Biological: Trivalent Invasive Salmonella Disease Vaccine (highest, well-tolerated dose among Cohorts A-C); Other: Placebo

INTERVENTIONS:
Biological: Trivalent Invasive Salmonella Disease Vaccine (6.25 µg) — 6.25 µg of the conjugate vaccine is administered via one intramuscular injection into the deltoid muscle on Study Day 1.
  Arms: Cohort A (Step 1)
Biological: Trivalent Invasive Salmonella Disease Vaccine (12 µg) — 12 µg of the conjugate vaccine is administered via one intramuscular injection into the deltoid muscle on Study Day 1.
  Arms: Cohort B (Step 2)
Biological: Trivalent Invasive Salmonella Disease Vaccine (25 µg) — 25 µg of the conjugate vaccine is administered via one intramuscular injection into the deltoid muscle on Study Day 1.
  Arms: Cohort C (Step 3)
Biological: Trivalent Invasive Salmonella Disease Vaccine (highest, well-tolerated dose among Cohorts A-C) — The highest, well-tolerated dose of the conjugate vaccine among Cohorts A-C is administered via one or two intramuscular injection(s) into the deltoid muscle on Study Day 1 (and 29 if two doses are given).
  Arms: Cohort D
Other: Placebo — 0.5 mL of buffer and preservative is administered via one or two intramuscular injections(s) into the deltoid muscle on Study Day 1 (and 29 if two doses are given).

SUMMARY:
This is a randomized, placebo-controlled dose-escalation study. The main purpose of this research is to test the safety and measure the immune response of the trivalent vaccine against invasive Salmonella disease. The vaccine will be tested over a range of doses.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Age 18 - 45 years, inclusive
* Good general health as determined by: vital signs (heart rate <100 bpm; blood pressure systolic >90 mm Hg and ≤150 mm Hg; diastolic >45 mm Hg and ≤90 mm Hg; oral temperature <100.4ºF), medical history, and a physical examination† within 45 days before administration of first dose of vaccine.
* Expressed interest and availability to fulfill the study requirements
* For females of child-bearing potential*, must agree to acceptable birth control&, 4 weeks before enrollment and through 4 weeks after last vaccination.
* Agrees not to participate in another clinical trial at any time during the study period.
* Agrees to allow for the indefinite storage of blood samples for future research use.

Exclusion Criteria:

* History of typhoid vaccination or known history of typhoid infection within 5 years
* Unacceptable laboratory abnormality from screening (prior to first vaccination) or upon safety laboratory testing (prior to second vaccination) as listed below. Laboratories with abnormalities which are possibly transient in nature may be repeated one time.

  1. Hemoglobin, white blood cell (WBC) count, absolute neutrophil count (ANC), or platelet count of an unacceptable value, according to Appendix B
  2. Creatinine, AST, ALT, total bilirubin, or C-reactive protein of an unacceptable value, according to Appendix B
  3. Positive serology for hepatitis C or HIV antibody or hepatitis B surface antigen.

(Subjects will be informed if their results are positive for hepatitis C, HIV antibody or hepatitis B surface antigen and will be referred to a primary care provider for follow up of these abnormal laboratory tests.)

* For women of child-bearing potential, positive serum pregnancy test (during screening within 45 days of enrollment) or positive urine pregnancy test (prior to and within 24 hours of administering each dose of vaccine).
* Nursing mother.
* Temperature > 38.0°C (100.4°F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 3 days prior to each dose of vaccine.
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* Diagnosis of schizophrenia or other major psychiatric disease
* Failure to pass Comprehension Assessment Tool during screening (70% correct answers are required to pass).
* Receipt of an experimental agent (vaccine, drug, device, etc.) within 28 days before enrollment or expects to receive an experimental agent during the study period.
* Receipt of any licensed vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) before enrollment in this study.
* Known sensitivity to any ingredient in the study vaccine, including a history of severe allergic reaction to tetanus vaccine.
* Receipt of immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Long-term use (>2 weeks) of oral or parenteral steroids (glucocorticoids), or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Frequency and Severity of Solicited Local and Systemic AEs | Approximately one year
  To assess the frequency and severity of solicited local (i.e., injective site) and systemic (such as fever) AEs during the first 7 days following each dose of vaccine.
Frequency and Severity of Unsolicited AEs and SAEs | Approximately two years
  To assess the frequency and severity of unsolicited AEs within 28 days of each dose of vaccine and the occurrence of any SAEs through 6 months after the last dose of vaccine
Proportion of Responders | Approximately one and a half years
  To measure the proportion of subjects that achieve a four-fold increase in titer, as compared to baseline, of specific serum IgG anti-COPS (S. Enteritidis or S. Typhimurium), anti-Vi (S. Typhi) polysaccharide, and anti-FliC (S. Enteritidis or S. Typhimurium) antibody at days 29 and 57, as measured by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen WH, Barnes RS, Sikorski MJ, Datar R, Sukhavasi R, Liang Y, Rapaka RR, Pasetti MF, Sztein MB, Wahid R, Tennant SM, Simon R, Baliban SM, Galen JE, Lees A, Bernshtein B, Alter G, Ella R, Mohan K, Naidu MG, Rao DY, Ella KM, Levine MM. A combination typhoid and non-typhoidal Salmonella polysaccharide conjugate vaccine in healthy adults: a randomized, placebo-controlled phase 1 trial. Nat Med. 2025 Dec;31(12):4256-4264. doi: 10.1038/s41591-025-04003-z. Epub 2025 Oct 8. PMID 41062830
- [Derived] Chen WH, Barnes RS, Sikorski MJ, Datar R, Sukhavasi R, Liang Y, Rapaka RR, Pasetti MF, Sztein MB, Wahid R, Tennant SM, Simon R, Baliban SM, Galen JE, Lees A, Bernshtein B, Alter G, Ella R, Mohan K, Naidu MG, Rao DY, Ella KM, Levine MM. A phase 1 randomized, placebo-controlled trial of a combination typhoid and non-typhoidal Salmonella polysaccharide conjugate vaccine. medRxiv [Preprint]. 2025 Sep 18:2025.09.15.25335795. doi: 10.1101/2025.09.15.25335795. PMID 41001453

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT03981952/Prot_SAP_000.pdf